CLINICAL TRIAL: NCT00374127
Title: Comparison Between Marijuana Smoked in Cigarette Paper (Joints) Versus Cigar Paper (Blunts)
Brief Title: Comparison Between Marijuana Smoked in Cigarette Paper Versus Cigar Paper
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 4683
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-07

CONDITIONS: Marijuana Dependence
Keywords: Marijuana; Comparison between joints and blunts; Pharmacokinetic effects
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- marijuana blunt (Experimental): marijuana blunt (0%, 1.8%, or 3.6% THC)
  Interventions: Drug: Marijuana blunt
- marijuana cigarette (Experimental): marijuana cigarette (0%, 1.8%, or 3.6% THC)
  Interventions: Drug: marijuana cigarette

INTERVENTIONS:
Drug: Marijuana blunt — Blunts were fabricated by cutting the bottom third off a Dutch Master® cigar, removing all of the cigar tobacco, and replacing it with all of the marijuana contained in a NIDA marijuana cigarette (ca. 800 mg).
  Other Names: Blunt
  Arms: marijuana blunt
Drug: marijuana cigarette — Marijuana cigarettes were provided by the National Institute on Drug Abuse.
  Other Names: Joint
  Arms: marijuana cigarette

SUMMARY:
The purpose of this study is to investigate whether or not marijuana blunts will produce comparable plasma THC levels as marijuana joints and if blunts will produce larger cardiovascular and subjective effects.

DETAILED DESCRIPTION:
There has been a rapid increase in marijuana use during the 1990s, with the most recent generation often smoking marijuana in the form of 'blunts' as opposed to more traditional routes such as in pipes or in cigarette paper. A blunt is made by removing the tobacco from a cigar and replacing it with marijuana (Golub and Johnson, 1999). The cigar wrapper contains tobacco and nicotine, which may interact with the cardiovascular and subjective effects of the marijuana to produce a different set of effects and risks than cigarette paper. Anecdotally, marijuana smokers report that blunts are more potent than joints, yet there have been no controlled studies addressing whether blunts enhance the subjective-effects and health-related consequences of marijuana use. We are proposing to do a within-subject, placebo-controlled study directly comparing the cardiovascular, subjective and pharmacokinetic effects of marijuana smoked in blunts compared to identical quantities of marijuana smoked in cigarette paper. Research volunteers will be current blunt smokers. Each will participate in six, 4-hour outpatient sessions. After baseline data have been collected (heart rate, blood pressure, mood scales, exhaled carbon monoxide, plasma THC and nicotine levels), participants will take 3 puffs, 5 seconds in duration, from a NIDA marijuana cigarette containing 0.0, 1.8 and 3.6% THC or from a blunt containing an equivalent quantity and strength of marijuana. Participants will be blind to the type of marijuana cigarette smoked. We will measure plasma THC and nicotine, subjective mood ratings, and heart rate and blood pressure repeatedly over the course of 180 minutes following smoking. This study is the first controlled investigation of the consequences of this new method of marijuana smoking; the data obtained may be useful in guiding future development of marijuana pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Current blunt marijuana use (minimum of twice/week) drug screen
* 21-45 years of age
* Practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD)

Exclusion Criteria:

* Current, repeated illicit drug use(excluding marijuana)
* Heavy cigarette use (> 10 cigarettes/day)
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease, hypertension)
* Laboratory tests outside normal limits that are clinically unacceptable to the study physician (BP > 140/90; hematocrit < 34 for women, < 36 for men)
* Significant adverse reaction to marijuana
* Current parole or probation
* Pregnancy or current lactation
* History of significant violent behavior
* Major current Axis I psychopathology(e.g., mood disorder with functional impairment or suicide risk, anxiety disorder, schizophrenia)
* History of heart disease
* Current use of any over-the-counter or prescription

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2004-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal, healthy volunteers ages 21-45 were recruited through newspaper advertisements and those who met inclusion/exclusion criteria after an initial phone screen were invited to the laboratory for further screening.
Pre-assignment Details: Prior to enrollment, participants gave written informed consent, received a psychiatric and medical evaluation, and provided a detailed drug use and medical history.
Groups:
- Marijuana: marijuana blunt (0%, 1.8%, or 3.6% THC) vs. marijuana cigarette (0%, 1.8%, or 3.6% THC)
Period: Overall Study
Arm/Group | Marijuana
Started | 35
Completed | 24
Not Completed | 11
Not completed — Did not inhale during smoking procedure. | 3
Not completed — Blood could not be drawn. | 2
Not completed — Protocol Violation | 5
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Marijuana
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.5 [21 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Plasma THC
Description: Plasma THC levels were analyzed to determine pharmacokinetic differences between marijuana cigarettes vs marijuana blunts.
Time Frame: 180 minutes
Population: Twenty four participants were included in this within-subjects analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Marijuana Blunt 0% THC: One of six within-subjects conditions where patients received a marijuana blunt containing 0% THC.
- Marijuana Blunt 1.8% THC: One of six within-subjects conditions where patients received a marijuana blunt containing 1.8% THC.
- Marijuana Blunt 3.6% THC: One of six within-subjects conditions where patients received a marijuana blunt containing 3.6% THC.
- Marijuana Cigarette 0% THC: One of six within-subjects conditions where patients received a marijuana cigarette containing 0% THC.
- Marijuana Cigarette 1.8% THC: One of six within-subjects conditions where patients received a marijuana cigarette containing 1.8% THC.
- Marijuana Cigarette 3.6% THC: One of six within-subjects conditions where patients received a marijuana cigarette containing 3.6% THC.
Arm/Group | Marijuana Blunt 0% THC | Marijuana Blunt 1.8% THC | Marijuana Blunt 3.6% THC | Marijuana Cigarette 0% THC | Marijuana Cigarette 1.8% THC | Marijuana Cigarette 3.6% THC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
ng/mL | 6 (1) | 53 (2) | 70 (2) | 7 (1) | 80 (3) | 98 (3)

2. Secondary Outcome: Subjective Effects on MRF
Description: Using the Marijuana Rating Form (MRF), subjective effects of "Take Again", "Liking", and "Strong" were assessed. The MRF is a visual analog scale allowing patients to indicate how they feel on a 100-mm line anchored with 'not at all' at the left end and 'extremely' at the right end, when prompted by a statement.
Time Frame: 180 minutes
Population: Twenty four participants were included in this within-subjects analysis.
Measure: Mean (Standard Deviation); unit: Ratings (mm)
Arm/Group | Marijuana Blunt 0% THC | Marijuana Blunt 1.8% THC | Marijuana Blunt 3.6% THC | Marijuana Cigarette 0% THC | Marijuana Cigarette 1.8% THC | Marijuana Cigarette 3.6% THC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Ratings (mm)
  "Take Again" | 23 (0.5) | 28 (0.4) | 36 (0.5) | 12 (0.4) | 45 (0.5) | 54 (0.4)
  "Liking" | 18 (0.4) | 30 (0.5) | 33 (0.4) | 10 (0.5) | 45 (0.4) | 55 (0.5)
  "Strong" | 10 (0.5) | 17 (0.4) | 29 (0.5) | 5 (0.4) | 30 (0.5) | 42 (0.4)

3. Secondary Outcome: Subjective Effects on VAS
Description: Subjective VAS ratings of 'Good Drug Effect' and 'High' averaged across all post-smoking time points when marijuana was smoked as joints and blunts analyzed for all participants. Here, participants indicated how they were feeling on a 100-mm line anchored with 'not at all' at the left end and 'extremely' at the right end, when prompted by a statement
Time Frame: 180 minutes
Population: Twenty-four participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: Ratings (mm)
Arm/Group | Marijuana Blunt 0% THC | Marijuana Blunt 1.8% THC | Marijuana Blunt 3.6% THC | Marijuana Cigarette 0% THC | Marijuana Cigarette 1.8% THC | Marijuana Cigarette 3.6% THC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Ratings (mm)
  Good Drug Effect | 10 (0.5) | 29 (0.4) | 33 (0.5) | 4 (0.4) | 28 (0.5) | 37 (0.4)
  High | 7 (0.4) | 10 (0.5) | 20 (0.4) | 3 (0.5) | 23 (0.4) | 30 (0.5)

4. Secondary Outcome: Carbon Monoxide
Description: Expired carbon monoxide averaged across all post-smoking time points when marijuana was smoked as joints and blunts for all participants.
Time Frame: 180 minutes
Population: Twenty-four participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Marijuana Blunt 0% THC | Marijuana Blunt 1.8% THC | Marijuana Blunt 3.6% THC | Marijuana Cigarette 0% THC | Marijuana Cigarette 1.8% THC | Marijuana Cigarette 3.6% THC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
ppm | 5.9 (0.5) | 6.4 (0.4) | 5.8 (0.5) | 5.5 (0.4) | 5.9 (0.5) | 5.3 (0.4)

5. Secondary Outcome: Heart Rate
Description: Heart rate averaged across all post-smoking time points when marijuana was smoked as joints and blunts.
Time Frame: 180 minutes
Population: Twenty-four participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Marijuana Blunt 0% THC | Marijuana Blunt 1.8% THC | Marijuana Blunt 3.6% THC | Marijuana Cigarette 0% THC | Marijuana Cigarette 1.8% THC | Marijuana Cigarette 3.6% THC
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
BPM | 70.5 (0.5) | 72.5 (0.4) | 73 (0.5) | 70.5 (0.4) | 72 (0.5) | 74 (0.4)

ADVERSE EVENTS:
Groups:
- Marijuana Blunt: marijuana blunt (0%, 1.8%, or 3.6% THC)
  Marijuana blunt
- Marijuana Cigarette: marijuana cigarette (0%, 1.8%, or 3.6% THC)
  marijuana cigarette
Arm/Group | Marijuana Blunt | Marijuana Cigarette
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
It is unknown if the cigar paper would provide physiologically relevant nicotine plasma levels under more extended durations of smoking. The small sample size prohibited an analysis to verify a statistically significant sex difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No